CLINICAL TRIAL: NCT05293691
Title: Body, Breath & Mind - A Randomized Control Trial to Test the Efficacy of an Online Self-help Program for Negative Affect and Depression
Brief Title: Efficacy of an Online Self-help Program for Negative Affect and Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Body, Breath & Mind
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Depressive Symptoms; Depression
Keywords: depression; quality of life; online; self-help program; randomized control trial; QiGong
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Body, Breath & Mind (Experimental): The program "Body, Breath & Mind" is a minimally guided self-help program to improve mood. It contains a total of eight modules, which are to be completed in a weekly rhythm. Each module includes Qi Gong exercises, and instructions and exercises for value-based behavioral activation used in behavioral therapy for depression (Hofheinz, Heidenreich & Michalak, 2017). If possible, the entire program should be completed within a period of 8 weeks.
  Interventions: Behavioral: Body, Breath & Mind
- Moodgym (Active Comparator): Moodgym is an interactive training program for the prevention and reduction of depressive symptoms. It is based on the methods and techniques of cognitive behavioral therapy and includes five modules: feelings, thoughts, developing alternative thoughts, deal with stress and relationship. In addition to the modules, there is a workbook section where personal results and responses are stored.The effectiveness of the programme has been proven in clinical trials (Loebner et al., 2018).
  Interventions: Behavioral: Moodgym
- Waitlist control group (Other): Participants in the waitlist control group are given access to the Body, Breath & Mind program after eight weeks, provided they have participated in the previous surveys in the form of a diagnostic pre-, peri-, and post-module.
  Interventions: Behavioral: Body, Breath & Mind

INTERVENTIONS:
Behavioral: Body, Breath & Mind — The program "Body, Breath & Mind" is a minimally guided self-help program to improve mood. It contains a total of eight modules, which are to be completed in a weekly rhythm. Each module includes Qi Gong exercises, and instructions and exercises for value-based behavioral activation used in behavioral therapy for depression (Hofheinz, Heidenreich & Michalak, 2017). If possible, the entire program should be completed within a period of 8 weeks.
  Arms: Body, Breath & Mind; Waitlist control group
Behavioral: Moodgym — Moodgym is an interactive training program for the prevention and reduction of depressive symptoms. It is based on the methods and techniques of cognitive behavioral therapy and includes five modules: feelings, thoughts, developing alternative thoughts, deal with stress and relationship. In addition to the modules, there is a workbook section where personal results and responses are stored. The effectiveness of the programme has been proven in clinical trials (Loebner et al., 2018).
  Arms: Moodgym

SUMMARY:
The aim of the study is to test Body, breath & mind (BBM, internet-based self-help program) for its efficacy in reducing depressive symptoms and improving quality of life. BBM combines methods of value-oriented behavioral activation with exercises from the Chinese healing practice Qi Gong,. BBM will be compared to an active control treatment (moodgym) and a waiting list control group. We expect significant differences to the waiting list control group. In comparison to the active control treatment we expect no significant differences.

ELIGIBILITY:
Inclusion Criteria:

* All persons who suffer from depressive symptoms (subthreshold and clinical depression; PHQ-9 ≥10)
* German speaking
* Internet and email access

Exclusion Criteria:

* The DSM-defined criteria A9 acute suicidality and A5 psychomotor agitation in the context of a depressive disorder, verified using the Diagnostic Interview in Mental Disorders in form of the Mini-DIPS (Margraf & Cwik, 2017)
* psychotic disorders, verified using the Diagnostic Interview in Mental Disorders in form of the Mini-DIPS (Margraf & Cwik, 2017)
* major depression with psychotic features, verified using the Diagnostic Interview in Mental Disorders in form of the Mini-DIPS (Margraf & Cwik, 2017)
* eating disorders, verified using the Diagnostic Interview in Mental Disorders in form of the Mini-DIPS (Margraf & Cwik, 2017)
* current or past schizo-affective disorder, verified using the Diagnostic Interview in Mental Disorders in form of the Mini-DIPS (Margraf & Cwik, 2017)
* current substance use disorder, verified using the Diagnostic Interview in Mental Disorders in form of the Mini-DIPS (Margraf & Cwik, 2017)
* inability to participate in the program due to physical, practical, or other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Brief Patient Health Questionnaire (PHQ-9) | Post-Measurement after 8 weeks
  Depression

SECONDARY OUTCOMES:
Short Form (36) Health Survey | Post-Measurement after 8 weeks
  Quality of life
Brief Patient Health Questionnaire (PHQ-9) | 6-Month-Follow-Up
  Depression

CONTACTS AND LOCATIONS:
Locations (1):
- Private Universität WItten/Herdecke, Witten, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lobner M, Pabst A, Stein J, Dorow M, Matschinger H, Luppa M, Maross A, Kersting A, Konig HH, Riedel-Heller SG. Computerized cognitive behavior therapy for patients with mild to moderately severe depression in primary care: A pragmatic cluster randomized controlled trial (@ktiv). J Affect Disord. 2018 Oct 1;238:317-326. doi: 10.1016/j.jad.2018.06.008. Epub 2018 Jun 5. PMID 29902736
- [Background] Hofheinz C, Heidenreich T, & Michalak J. Werteorientierte Verhaltensaktivierung bei depressiven St rungen: Therapiemanual: mit E-Book inside und Arbeitsmaterial. Beltz. 2017.
- [Background] Margraf J, Cwik CC, Pflug V & Schneider S. Structured clinical interviews for mental disorders across the lifespan: Psychometric quality and further developments of the DIPS Open Access interviews. Zeitschrift für Klinische Psychologie und Psychotherapie. 2017; 46(3), 176-186.